CLINICAL TRIAL: NCT01109329
Title: Phase 1 Inpatient Study of rHMPV-SHs, a Human Metapneumovirus Challenge Strain, Administered to Healthy Adults in Isolation
Brief Title: Safety Study of a Human Metapneumovirus Challenge Virus in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CIR 270
Record Dates: First submitted 2010-04-21; First posted 2010-04-23 (Estimated); Last update posted 2013-01-03 (Estimated); Status verified 2012-12

CONDITIONS: Human Metapneumovirus
Keywords: Vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- HMPV challenge virus (Experimental): Participants will receive the HMPV challenge virus.
  Interventions: Biological: HMPV challenge virus

INTERVENTIONS:
Biological: HMPV challenge virus — Single dose of 10^6 plaque forming units (PFU) of recombinant HMPV small hydrophobic genes (rHMPV-SHs)

SUMMARY:
Human metapneumovirus (HMPV) is a virus that can cause respiratory illness. In older adults, those with asthma, infants, and children, illness can be severe, but in healthy adults the virus frequently causes no symptoms. The National Institute of Allergy and Infectious Diseases (NIAID) is working to develop a vaccine for HMPV that could be given to infants. Before potential vaccines can be tested, information about how HMPV affects healthy adults is needed. This study will examine the effects of exposure to HMPV in healthy adults.

DETAILED DESCRIPTION:
Human metapneumovirus (HMPV), a virus that causes respiratory illness, was first discovered in 2001, although humans have been infected with it for at least 50 years. HMPV may cause upper respiratory illness or no symptoms at all in healthy adults, but older adults, adults with asthma, and children may be at risk of more serious illness. HMPV is a leading cause of viral lower respiratory infection (LRI) in children, so finding a vaccine for this virus could substantially reduce the instances of childhood respiratory illnesses.

The National Institute of Allergy and Infectious Diseases (NIAID) is developing a vaccine for HMPV for use in infants, but before starting clinical trials with potential HMPV vaccines, researchers need to study how wild HMPV affects healthy adults. This study will expose healthy adults to a dose of the HMPV virus to assess its ability to infect, cause disease, and create an immune system response.

Participation in this study will last approximately 6 months. Participants will be admitted to an inpatient unit, where they will stay for 10 full days. On their second day in the unit, participants will receive a single dose of the virus, delivered via nose drops. Twice each day while participants are inpatients, they will undergo physical exams and have their vital signs recorded. Nasal washes and blood samples will be collected before participants receive the virus, and then daily nasal washes will be collected until they are discharged from the inpatient unit. Participants will be discharged from the unit on the 9th day after receiving virus if their nasal wash from Day 8 was free of virus. Follow-up visits will occur 28, 120, and 180 days after participants receive the virus. During follow-up visits nasal washes and blood samples will be collected.

ELIGIBILITY:
Inclusion Criteria:

* General good health, without significant medical illness, physical examination findings, or significant laboratory abnormalities as determined by the investigator
* Available for the duration of the trial
* Female subjects must agree to use effective birth control methods for the duration of the study

Exclusion Criteria:

* Pregnant
* Currently breastfeeding
* Evidence of clinically significant diseases in the nervous system, heart, lungs, liver, autoimmune system, or kidney or involving rheumatism, as determined by medical history, physical examination, or laboratory studies, including urine testing.
* Clinically significant alanine aminotransferase (ALT) levels, as determined by the principal investigator (PI)
* Behavioral or cognitive impairment or psychiatric disease that, in the opinion of the investigator, affects the ability to understand and cooperate with the study protocol
* Human metapneumovirus (HMPV) specific serum immunoglobulin A (IgA) titer greater than 1:50
* HMPV-specific nasal wash IgA titer greater than 1:50
* Positive urine drug toxicology test indicating narcotic use
* Medical, occupational, or family problems as a result of alcohol or illicit drug use during the past 12 months
* Other condition that, in the opinion of the investigator, would jeopardize the safety or rights of a subject participating in the trial or would render the subject unable to comply with the protocol
* History of hypersensitivity reactions
* Diagnosis of asthma or reactive airway disease within the past 2 years
* Positive result on test for HIV
* Positive result on test for hepatitis C virus (HCV)
* Positive result on test for hepatitis B virus surface antigen (HBsAg)
* Known immunodeficiency syndrome
* Use of corticosteroids (excluding topical or nasal preparations) or immunosuppressive drugs within 30 days prior to inoculation
* Receipt of a live vaccine within 4 weeks or a killed vaccine within 2 weeks prior to inoculation with challenge virus, rHMPV-SHs
* History of a surgical removal of the spleen
* Receipt of blood or blood-derived products (including immunoglobulin) within 6 months prior to study inoculation
* Current smoker unwilling to stop smoking for the duration of the study
* Receipt of another investigational vaccine or drug within 30 days prior to study inoculation
* Body mass index (BMI) greater than 35
* Shares household with a child younger than 60 months of age or an immunocompromised individual
* Unwillingness to have nasal wash or blood samples saved for future respiratory virus research

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2010-06; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Frequency of challenge virus (rHMPV-SHs) infection, defined as virus shedding in respiratory secretions or serological evidence of HMPV infection | Measured at baseline and on Days 1 to 9
rHMPV-SHs shedding, as measured by peak virus titer, mean sum of daily virus titers, and total duration of shedding | Measured at baseline and on Days 1 to 9
Frequency and severity of respiratory illness | Measured at study completion

SECONDARY OUTCOMES:
Magnitude, frequency, and duration of serum and nasal wash antibody responses induced by rHMPV-SHs | Measured at baseline and on Days 28, 120, and 180
Correlation between virus shedding and severity of clinical illness | Measured at study completion
Cytokine and chemokine concentrations in nasal wash samples and relationships between cytokine/chemokine induction, viral replication, and illness | Measured at study completion
T-cell mediated and innate immune responses | Measured at baseline and on Days 8, 28, and 180
Whether HMPV infection induces characteristic gene expression patterns in cells obtained from blood or nasal wash | Measured at baseline and Days 3, 5, 7, 8, 28, and 180
Relationship between the development of immune responses and clearance of rHMPV-SHs | Measured at study completion

CONTACTS AND LOCATIONS:
Overall Officials: Ruth Karron, MD, Principal Investigator — Johns Hopkins University, Bloomberg School of Public Health
Locations (1):
- Johns Hopkins Bloomberg School of Public Health, Baltimore, Maryland, United States

REFERENCES:
- [Background] Bruno R, Marsico S, Minini C, Apostoli P, Fiorentini S, Caruso A. Human metapneumovirus infection in a cohort of young asymptomatic subjects. New Microbiol. 2009 Jul;32(3):297-301. PMID 19845113
- [Background] Williams JV, Harris PA, Tollefson SJ, Halburnt-Rush LL, Pingsterhaus JM, Edwards KM, Wright PF, Crowe JE Jr. Human metapneumovirus and lower respiratory tract disease in otherwise healthy infants and children. N Engl J Med. 2004 Jan 29;350(5):443-50. doi: 10.1056/NEJMoa025472. PMID 14749452
- [Derived] Talaat KR, Luke CJ, Khurana S, Manischewitz J, King LR, McMahon BA, Karron RA, Lewis KD, Qin J, Follmann DA, Golding H, Neuzil KM, Subbarao K. A live attenuated influenza A(H5N1) vaccine induces long-term immunity in the absence of a primary antibody response. J Infect Dis. 2014 Jun 15;209(12):1860-9. doi: 10.1093/infdis/jiu123. Epub 2014 Mar 5. PMID 24604819
- [Derived] Talaat KR, Karron RA, Thumar B, McMahon BA, Schmidt AC, Collins PL, Buchholz UJ. Experimental infection of adults with recombinant wild-type human metapneumovirus. J Infect Dis. 2013 Nov 15;208(10):1669-78. doi: 10.1093/infdis/jit356. Epub 2013 Aug 1. PMID 23908489